CLINICAL TRIAL: NCT05987176
Title: An International Multicentre Randomized Unblinded Phase II Study Comparing Adjuvant Treatment With 177Lu-DOTATATE (Lutathera®) to Best Supportive Care in Patients After Resection of Neuroendocrine Liver Metastases
Brief Title: Comparison of Adjuvant Treatment With 177Lu-DOTATATE to Best Supportive Care in Patients After Resection of Neuroendocrine Liver Metastases
Acronym: NELMAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has closed earlier than planned due to one of the funders decision to withdraw the financial support for the study.
Sponsor: Imperial College London (Other)
Collaborators: The Taylor Family 2010 Charitable Trust (Unknown); Novartis/AAA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF-ICL 01; 2022-003575-42 (EudraCT Number)
Record Dates: First submitted 2023-03-08; First posted 2023-08-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Neuroendocrine Tumor G1 (NET G1)/Carcinoid; Neuroendocrine Tumor Grade 2; Neuroendocrine Tumors; Liver Metastases; Gastroenteropancreatic Neuroendocrine Tumor; Gastroenteropancreatic Neuroendocrine Neoplasm
Keywords: NETs; NECs; GEP-NETs; NELMAS; adjuvant; liver metastases
MeSH Terms: conditions — Neuroendocrine Tumors; Gastro-enteropancreatic neuroendocrine tumor | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care - Arm A (No Intervention): Control arm as per standard of care patients go on routine follow up post surgery.
  The control arm will consist of best supportive care. The study will be embedded within the regular clinical pathway for treatment and follow-up of patients with resectable NE LM. The follow-up will be according to current guidelines (e.g., Guidelines of the European Neuroendocrine Tumor Society for the management of advanced intestinal NET and pancreatic NET with locoregional and/or distant metastases).
  Patients will be followed up in the study for 3 years according to standard post-surgical follow-up protocol and thereafter in their local institution life-long according to follow-up after liver resection for NE LM
- Treatment - Arm B (Experimental): Treatment with Lutathera post surgery.
  In the treatment arm 177Lu-DOTATATE will be applied. The frequency of administration will be 2 cycles (8±1weeks between each cycle). The rationale for 2 cycles instead of 4 (as per standard protocol in palliative setting), assumes that there will be no macroscopic residual tumour after liver resection. Thus, the treatment dose should be sufficient to target microscopic disease, and at the same time have smallest possible effect on healthy tissue.
  Interventions: Drug: Lutathera

INTERVENTIONS:
Drug: Lutathera — Dosage:
  In total 14.8 GBq (400 mCi) 177Lu-DOTATATE administered in two equally divided doses. Each dose to be infused over 30 minutes.
  Duration of treatment:
  Two administrations of 177Lu-DOTATATE (each treatment 7.4 GBQ (200 mCi) at 8±1-week intervals, which can be extended to 16 weeks for resolving acute toxicity.
  Arms: Treatment - Arm B

SUMMARY:
An international multi-centre, open, randomised, parallel-group phase II study comparing adjuvant treatment with 177Lu-DOTATATE to best supportive care in patients after complete surgical removal of neuroendocrine liver metastases.

In this study, adjuvant treatment with 177Lu-DOTATATE will be compared with best supportive care in patients with well differentiated grade 1 or 2 neuroendocrine tumours in the stomach, pancreas or gut (gastro-entero-pancreatic NETs) who had their primary tumour already removed or in whom both primary and liver tumour metastases removal will take place simultaneously, including removal of perihilar lymph nodes will be eligible.

The primary objective is to compare overall disease-free survival at 3 years after treatment with 177Lu-DOTATATE to best supportive care between both treatment arms, with equal chances of entering either arm (1:1)

Secondary objectives are to describe and compare the difference in disease-free survival in the liver, overall survival, time to the next anticancer treatment, the cost effectiveness and health-related quality of life. The safety and toxicity of 177Lu-DOTATATE as adjuvant therapy will also be described.

Additionally, the clinical use of blood and urine analysis test (NETest) will be evaluated to identify microscopic remaining disease and detect early the return of the tumour.

DETAILED DESCRIPTION:
There will be 2 arms: arm A consisting of best supportive care and arm B, the experimental treatment. Randomisation will be 1:1 as soon as possible after the liver surgery.

The control arm will consist of standard of care. The study will be embedded within the regular clinical pathway for treatment and follow-up of patients with resectable NE LM. The follow-up will be according to current guidelines (e.g., Guidelines of the European Neuroendocrine Tumor Society for the management of advanced intestinal NET and pancreatic NET with locoregional and/or distant metastases). Patients will be followed up in the study for 3 years according to standard post-surgical follow-up protocol and thereafter in their local institution life-long according to follow-up after liver resection for NE LM.

In the treatment arm 177Lu-DOTATATE will be applied. The first cycle will be applied 6±2 weeks after liver resection. The frequency of administration will be 2 cycles (8±1weeks between each cycle). The rationale for 2 cycles in the adjuvant setting instead of 4 (as per standard protocol in palliative setting), assumes that after the removal of the primary tumour and the liver metastases, there will be no macroscopic residual tumour. Thus, the treatment dose should be sufficient to target microscopic disease and have the smallest possible effect on healthy tissue.

In the treatment arm, the patients will have 10 study visits for post -PRRT monitoring (blood tests and clinical assessments). Patients in the standard of care arm will have visits every 3 months. In both arms, patients will have one screening visit and one end of study visit. They will complete QoL questionnaires at baseline and at follow-up visits at 12, 24, and 36 months and bloods/urine will be collected for translational research prior to surgery (while in hospital) and at 6, 12, and 36 months.

Signature of informed consent precedes all study-specific assessments. All patients will have a fresh tumour sample collected during the liver surgery. Disease recurrence will be measured in all patients using liver MRIs every 3 months for the first year and every 6 months for the second to third year and 68Ga DOTA-TATE PET CT every 12 months for 3 years. Any patient with disease recurrence ceases treatment and assessments and will proceed to standard of care treatment for recurrent liver metastases.

Follow-up data will be collected for 5 years overall from the date of randomisation of the last patient.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any study related procedures
2. Patients aged 18 years or older
3. ECOG / WHO performance status 0 or 1
4. Patients with well differentiated grade 1 or grade 2 (Ki67<20%) GEP NET confirmed by histological criteria with the primary localisation in stomach, pancreas, or gut
5. Patients after R0 (complete macroscopic and microscopic resection) or R1 (complete macroscopic resection, microscopically positive resection margins) resection of neuroendocrine liver metastases confirmed by histological criteria
6. Patients with a primary tumour already resected or in whom the primary tumour has been resected synchronously with liver metastases
7. MRI scan prior to surgery (within 4 -6 weeks) confirming liver metastases and no extrahepatic disease (except resectable perihilar lymph node involvement and/or primary tumour, if still in place)
8. Somatostatin receptor-based imaging (68Ga DOTA-TATE PET/CT prior to surgery (within 12 weeks) confirming liver metastases and no extrahepatic disease (except resectable perihilar lymph node involvement and/or primary tumour, if still in place)

Exclusion Criteria:

1. Less than 4 weeks post-surgery, or any other medical treatment, including chemotherapy, radiotherapy, and intrahepatic therapy
2. High grade neuroendocrine tumours (G3 NET, or neuroendocrine carcinoma [NEC])
3. After R2 (tumour debulking, macroscopically incomplete resection) resection of neuroendocrine liver metastases
4. Patients with non-resectable neuroendocrine liver metastases and/or non-resectable primary tumour and /or non-resectable perihilar lymph node metastases
5. Pregnancy
6. Subjects of childbearing potential (both male and female participants) not willing to use a combination of adequate contraceptive measures, e.g., oral contraceptives, IUD, barrier methods of contraception (condom or occlusive cap with spermicide)
7. Patients who have received prior systemic and/or liver-directed treatment for their metastatic NET other than somatostatin analogues
8. Hb concentration <5.0 mmol/L (<8.0 g/dL)
9. WBC <2x109/L (2000/mm3)
10. Platelets <75x109/L (75x103/mm3).
11. Total bilirubin >3 x ULN.
12. Serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
13. Uncontrolled congestive heart failure (NYHA II, III, IV).
14. Uncontrolled diabetes mellitus as defined by a fasting blood glucose >2 ULN.
15. Prior external beam radiation therapy to more than 25% of the bone marrow.
16. Kidney failure with serum creatinine >150 µmol/L (>1.7 mg/dL)
17. Known hypersensitivity to somatostatin analogues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 3 years
  To compare overall Disease-Free Survival (DFS) at 3 years after treatment with 177Lu-DOTATATE to best supportive care in patients with R0/R1 resected liver metastases of well differentiated (grade 1 or 2) GEP NET and no extrahepatic disease manifestation prior to randomization in the study.

SECONDARY OUTCOMES:
Comparison of Disease free survival in the liver between arm | 3 years
  To compare the Disease-Free Survival (DFS) in the liver between the two study arms
Overall survival | 5 years
  To compare the overall survival (OS) in the liver between the two study arms
Time to tumour recurrence | 5 years
  To compare the Time to Tumour Recurrence (TTR) between the two study arms
Comparison Time to next antineoplastic therapy | 5 years
  To compare the time to administration of subsequent antineoplastic therapy between the two arms
Safety and tolerability of 177Lu-DOTATATE (AEs/SAEs/SUSARs) | 5 years
  To evaluate the safety and tolerability of 177Lu-DOTATATE
Evaluation of quality of life | 3 years
  To evaluate the health-related Quality of Life (QoL) as measured by the EORTC QLQ-C30, QLQ-GI NET 2.1 and EQ-5D questionnaires
Evaluation of self reported health perceptions | 3 years
  To evaluate patient reported outcomes (PROs) as measured by the Short Form-36® (SF-36) Health Survey
Cost-effectiveness evaluation | 5 years
  To evaluate the cost effectiveness assessed by EuroQol-5D (cost for subsequent therapy)

OTHER OUTCOMES:
NETest | 3 years
  • To explore the clinical utility of novel biomarkers (NETest, PPQ, metabolic signature) in identification of residual microscopic disease and early detection of recurrent disease

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Frilling, Prof, Study Chair — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No